CLINICAL TRIAL: NCT05356962
Title: STOP? II Trial: Cluster Randomized Clinical Trial to Test the Implementation of a Toolbox for Structured Communication in the Operating Room
Brief Title: STOP? II: Testing of a Toolbox for Structured Communication in the Operating Room
Acronym: StOP?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); University of Bern (Other); Fachhochschule Nordwestschweiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021-02433
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Communication Research; Communication, Multidisciplinary
Keywords: Communication; Briefing; Intervention; Operating room; Surgery
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind whether the patients were operated by a surgeon in the control or in the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The surgeons will undergo a multi-module training on how to use the StOP?-protocol and perform the StOP?-protocol during all their operations during a 4-month period.
  Interventions: Behavioral: StOP?-protocol
- Control group (No Intervention): Surgeons in the control group will not be trained to the StOP?-protocol and will communicate as usual during their operations.

INTERVENTIONS:
Behavioral: StOP?-protocol — The StOP?-protocol is an intra-operative briefing initiated by the responsible surgeon. When performing a StOP?-protocol, the surgeons inform the team present in the operating room about the Status (St) of the operation, the Objectives (O) of the operations, the potential problems (P) they may meet and encourage the team to ask questions or voice concerns (?). The responsible surgeon announces at the team timeout when they plan to perform the StOP-protocol(s).
  Arms: Interventional group

SUMMARY:
The purpose of the study is to test the impact of the StOP?-protocol - an intra-operative communication briefing, on post-operative mortality and important patient outcomes.

DETAILED DESCRIPTION:
The StOP?-protocol is a communication briefing initiated by the responsible surgeon during a surgical operation. The surgeon informs the team present in the operating room about the current Status of the operation, the Objectives of the next steps and the potential Problems the surgical team may meet; the responsible surgeon encourages the team to voice any question or concern (?).

To test the impact of the StOP?-protocol on patient outcomes, the study is designed as a randomized controlled trial. Surgeons will be randomized either (a) in the intervention group and be trained to perform the StOP?-protocol or (b) in the control group and will communicate as they prefer during their operations. Post-operative patient outcomes of the surgeons in the intervention and the control group will be compared to evaluate the effects of the StOP?-protocol.

ELIGIBILITY:
For the clusters (surgeons)

Inclusion Criteria:

* Board-certified surgeons with specialization in one of the following disciplines: general, visceral, thoracic, vascular surgery, surgical urology, or gynecology.

Exclusion Criteria:

* Surgeons who are already performing StOP?-protocol. (Potentially, surgeons who took part in the first study (StOP-I) may still perform StOP?).
* Surgeon who were previously enrolled in the StOP?-II trial (this is relevant for surgeons who move or rotate between departments/hospitals and might therefore be working at different participating sites).

For the patients:

Inclusion criteria:

* Patients operated by cluster surgeons during the cluster-specific time period
* General consent from the patients, allowing the use of healthcare-related data that are the result of the patient's treatment. In case no written document from the general consent is available despite documented efforts of the participating center, article 34 HRA (Swiss law) will be applied, allowing the use of the healthcare-related patient data.

Exclusion criteria:

* Patient age below 18 years
* Previous operation at the same site up to 30 days prior the index operation
* Procedures not done in operating rooms but in outpatient clinics, on wards, etc.
* Mainly diagnostic endoscopic procedures (e.g. colonoscopy, gastroscopy, bronchoscopy)
* Percutaneous interventions (e.g., transurethral interventions)
* Documented refusal for the use of healthcare related data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Mortality within 30 days after the operation | 30 days after the index operation
  Mortality within 30 days after the operation in the intervention arm compared to the control arm

SECONDARY OUTCOMES:
Unplanned reoperations within 30 days after the operation | 30 days after the index operation
  Unplanned reoperations within 30 days after the operation in the intervention arm compared to the control arm
Length of hospital stay | It is reasonable to estimate that the information will be available after 60 post-operative days for most patients
  Length of hospital stay in the intervention arm compared to the control arm
Unplanned hospital readmissions within 30 days after the operation | 30 days after the index operation
  Unplanned hospital readmissions within 30 days after the operation in the intervention arm compared to the control arm

OTHER OUTCOMES:
Surgical site infections (SSI) within 30 days after the index operation | 30 days after the index operation
  Surgical site infections as defined by the Centers for Disease Control and Prevention (CDC) and collected by Swissnoso (a national surveillance programme for surgical site infections in Switzerland) in the intervention arm compared to the control arm. Note. SSI will be collected only for a pragmatic subsample of patients

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, MD, Principal Investigator — Department of Visceral Surgery and Medicine, Berne University Hospital, University of Berne, Berne, Switzerland
Locations (13):
- Tirol Kliniken GmbH, Innsbruck, Austria
- Switzerland (12):
  - Kantonsspital Baselland, Liestal, Basel-Landschaft
  - Kantonsspital Baden AG, Baden, Canton of Aargau
  - Bern University Hospital (Inselspital), Bern, Canton of Bern
  - Hôpital Fribourgeois, Fribourg, Canton of Fribourg
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Spital Limmattal, Schlieren, Canton of Zurich
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Stadtspital Zürich Triemli, Zurich, Canton of Zurich
  - EOC Civico Lugano and EOC ospedale regionale di Bellinzona, Lugano, Canton Ticino
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
  - Spital Thurgau, Frauenfeld, Thurgau
  - Réseau hospitalier neuchâtelois, Neuchâtel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Keller S, Tschan F, Semmer NK, Trelle S, Manser T, Beldi G. StOP? II trial: cluster randomized clinical trial to test the implementation of a toolbox for structured communication in the operating room-study protocol. Trials. 2022 Oct 18;23(1):878. doi: 10.1186/s13063-022-06775-y. PMID 36258223